CLINICAL TRIAL: NCT00166712
Title: A Phase IV, Single Center Pilot Study Using Alemtuzumab (Campath-1H) Induction Combined With Prednisone-Free, Calcineurin-Inhibitor-Free Immunosuppression in Kidney Transplantation
Brief Title: A Trial of Two Steroid-Free Approaches Toward Mycophenolate Mofetil-Based Monotherapy Immunosuppression
Acronym: Cell220
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study stopped due to lack of efficacy & funding.
Sponsor: Northwestern University (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Joseph Leventhal, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU8789 0811-007; CNV0042139 (Other Grant/Funding Number: Roche Laboratories, Inc.)
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Results first posted 2015-01-15 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Kidney Transplant Failure and Rejection
Keywords: Kidney Transplant; Living Donor Kidney Transplant Recipients
MeSH Terms: conditions — Rejection, Psychology | interventions — Tacrolimus; Sirolimus; Alemtuzumab; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: Alemtuzumab + TAC + MMF (Active Comparator): Receive two doses of alemtuzumab (Campath-1H, 30mg) by intravenous (IV) infusion. One dose during kidney transplant surgery and the second dose on day 2 (post-surgery) to achieve peripheral T-cell depletion. IV glucocorticoids will be given prior to Campath administration to limit cytokine release syndrome in association with this monoclonal antibody. MMF on the day of surgery and continue taking it by mouth, twice daily. TAC started on the 1st day after surgery, and then taken by mouth twice daily.
  Interventions: Drug: Tacrolimus (TAC); Drug: Alemtuzumab; Drug: Mycophenolate mofetil (MMF)
- Group 2: Alemtuzumab + Sirolimus + MMF (Active Comparator): Sirolimus will be taken by mouth before transplant surgery and will continue taking once daily after surgery. Group 2 will also receive 2 doses of Alemtuzumab: one during surgery and the second will be given on the second day after surgery. Mycophenolate mofetil will be give on the day of surgery and twice daily, by mouth, as instructed by the doctor.
  If subjects do not experience kidney rejection after 6 months after surgery, they will be weaned off of the sirolimus and continue taking the mycophenolate mofetil.
  Interventions: Drug: Sirolimus; Drug: Alemtuzumab; Drug: Mycophenolate mofetil (MMF)

INTERVENTIONS:
Drug: Tacrolimus (TAC) — Tacrolimus (TAC) will be given standard of care by prescription twice a day (2.0 mg), orally. Doses will be adjusted by serum levels. The dose will be modified to achieve 12 hour trough concentrations of 5-8 ng/mL.
  Other Names: Prograf®; FK506
  Arms: Group 1: Alemtuzumab + TAC + MMF
Drug: Sirolimus — Sirolimus will be given standard of care by prescription, dosed at 5mg daily. The dosage will be adjusted by serum level to achieve 24 hour trough concentrations of 8-12 ng/mL by HPLC assay.
  Other Names: Rapamune®; Rapamycin
  Arms: Group 2: Alemtuzumab + Sirolimus + MMF
Drug: Alemtuzumab — Patients receiving alemtuzumab will be premedicated with 50mg of diphenhydramine hydrochloride, and 650mg of acetaminophen 30-60 minutes to the first Alemtuzumab infusion. The of 30mg will be diluted in 100cc sterile 0.9% normal saline and infused over 2 hours. The infusion line must contain an in-line 0.22-micron filter. Alemtuzumab will be administered on the day of transplant (intraoperatively), and on post-operative day 2. Both doses will be administered while the patient is in the hospital. Alemtuzumab is supplied in single-use clear glass ampoules containing 30mg of alemtuzumab in 3mL of solution.
  Other Names: Campath®; Campath-1H; Mabcampath®
Drug: Mycophenolate mofetil (MMF) — MMF will be given at 1.0-1.5gm, twice daily, orally. The first dose will be given pre-transplant, open label fashion.
  Other Names: Cellcept®

SUMMARY:
This is an open label, single-center, randomized phase IV pilot study of steroid and calcineurin inhibitor avoidance in renal transplant recipients. All patients will receive two doses of alemtuzumab to achieve peripheral T-cell depletion. Intravenous glucocorticoids will be administered prior to alemtuzumab administration to limit cytokine release syndrome in association with this monoclonal antibody, and continued for the first two days post-transplant. Thereafter, steroids will not be used for immunosuppression. All transplant recipients will be started on oral immunosuppressive therapy with mycophenolate mofetil (MMF) prior to transplant. Pretransplant, these patients will be randomized to receive, in addition, either tacrolimus (Tac) or sirolimus.

After six months, patients in the tacrolimus arm who do not experience rejection will be randomized to continue on tacrolimus or to be converted to the combination of sirolimus and MMF. Individuals in this arm of the study who do not experience acute rejection, and demonstrate evidence of donor specific hyporesponsiveness at 9 months post-transplant (those staying on Tac + MMF) or 3 months post-conversion (those converted from Tac + MMF to sirolimus + MMF) will be weaned to MMF monotherapy.

Individuals in the sirolimus + MMF arm who do not experience acute rejection and demonstrate evidence of donor specific hyporesponsiveness at 6 months post-transplant will be weaned to MMF monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are male or female age 18-65 years
2. Donor age 18-65 years
3. Patients who are single-organ recipients (kidney only)
4. Women who are of childbearing potential must have a negative serum pregnancy test before transplantation and agree to use a medically acceptable method of contraception throughout the treatment period.
5. Subject (recipient) is able to understand the consent form and give written informed consent

Exclusion Criteria:

1. Known sensitivity or contraindication to sirolimus, tacrolimus or MMF
2. Patient with significant or active infection
3. Patients with a positive lymphocytotoxic crossmatch using donor lymphocytes and recipient serum
4. Patients with PRA > 20%
5. Patients who are pregnant or nursing mothers
6. Patients whose life expectancy is severely limited by diseases other than renal disease
7. Ongoing active substance abuse, drug or alcohol
8. Major ongoing psychiatric illness or recent history of noncompliance
9. Significant cardiovascular disease (e.g.):

   * Significant non-correctable coronary artery disease
   * Ejection fraction below 30%
   * History of recent myocardial infarction
10. Malignancy within 3 years, excluding non-melanoma skin cancers
11. Serologic evidence of infection with HIV or HBVsAg positive
12. Patients with a screening/baseline total white blood cell count < 4,000/mm3; platelet count < 100,000/mm3; triglycerides > 400 mg/dl; total cholesterol > 300 mg/dl
13. Investigational drug within 30 days prior to transplant surgery
14. Anti-T cell therapy within 30 days prior to transplant surgery
15. Patients using Prednisone
16. Patients who are ABO incompatible

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph R Leventhal, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University/Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Eggers PW. Effect of transplantation on the Medicare end-stage renal disease program. N Engl J Med. 1988 Jan 28;318(4):223-9. doi: 10.1056/NEJM198801283180406. PMID 3275896
- [Background] Hariharan S, Johnson CP, Bresnahan BA, Taranto SE, McIntosh MJ, Stablein D. Improved graft survival after renal transplantation in the United States, 1988 to 1996. N Engl J Med. 2000 Mar 2;342(9):605-12. doi: 10.1056/NEJM200003023420901. PMID 10699159
- [Background] Barry JM. Immunosuppressive drugs in renal transplantation. A review of the regimens. Drugs. 1992 Oct;44(4):554-66. doi: 10.2165/00003495-199244040-00003. PMID 1281071
- [Background] Suthanthiran M, Strom TB. Renal transplantation. N Engl J Med. 1994 Aug 11;331(6):365-76. doi: 10.1056/NEJM199408113310606. No abstract available. PMID 7832839
- [Background] Helderman JH, Van Buren DH, Amend WJ Jr, Pirsch JD. Chronic immunosuppression of the renal transplant patient. J Am Soc Nephrol. 1994 Feb;4(8 Suppl):S2-9. doi: 10.1681/ASN.V48s2. PMID 8193291
- [Background] Gaston RS. Maintenance immunosuppression in the renal transplant recipient: an overview. Am J Kidney Dis. 2001 Dec;38(6 Suppl 6):S25-35. doi: 10.1053/ajkd.2001.28923. PMID 11729003
- [Background] Pirsch JD, D'Alessandro AM, Sollinger HW, Knechtle SJ, Reed A, Kalayoglu M, Belzer FO. Hyperlipidemia and transplantation: etiologic factors and therapy. J Am Soc Nephrol. 1992 Jun;2(12 Suppl):S238-42. doi: 10.1681/ASN.V212s238. PMID 1498281
- [Background] Shaw LM, Kaplan B, Kaufman D. Toxic effects of immunosuppressive drugs: mechanisms and strategies for controlling them. Clin Chem. 1996 Aug;42(8 Pt 2):1316-21. PMID 8697605
- [Background] Boubenider S, Hiesse C, Goupy C, Kriaa F, Marchand S, Charpentier B. Incidence and consequences of post-transplantation lymphoproliferative disorders. J Nephrol. 1997 May-Jun;10(3):136-45. PMID 9238621
- [Background] Fishman JA, Rubin RH. Infection in organ-transplant recipients. N Engl J Med. 1998 Jun 11;338(24):1741-51. doi: 10.1056/NEJM199806113382407. No abstract available. PMID 9624195
- [Background] DeMario MD, Liebowitz DN. Lymphomas in the immunocompromised patient. Semin Oncol. 1998 Aug;25(4):492-502. PMID 9728599
- [Background] Sia IG, Paya CV. Infectious complications following renal transplantation. Surg Clin North Am. 1998 Feb;78(1):95-112. doi: 10.1016/s0039-6109(05)70637-x. PMID 9531938
- [Background] Pirsch JD, Miller J, Deierhoi MH, Vincenti F, Filo RS. A comparison of tacrolimus (FK506) and cyclosporine for immunosuppression after cadaveric renal transplantation. FK506 Kidney Transplant Study Group. Transplantation. 1997 Apr 15;63(7):977-83. doi: 10.1097/00007890-199704150-00013. PMID 9112351
- [Background] Ahsan N, Hricik D, Matas A, Rose S, Tomlanovich S, Wilkinson A, Ewell M, McIntosh M, Stablein D, Hodge E. Prednisone withdrawal in kidney transplant recipients on cyclosporine and mycophenolate mofetil--a prospective randomized study. Steroid Withdrawal Study Group. Transplantation. 1999 Dec 27;68(12):1865-74. doi: 10.1097/00007890-199912270-00009. PMID 10628766
- [Background] Vincenti F, Ramos E, Brattstrom C, Cho S, Ekberg H, Grinyo J, Johnson R, Kuypers D, Stuart F, Khanna A, Navarro M, Nashan B. Multicenter trial exploring calcineurin inhibitors avoidance in renal transplantation. Transplantation. 2001 May 15;71(9):1282-7. doi: 10.1097/00007890-200105150-00017. PMID 11397963
- [Background] Randhawa PS, Shapiro R, Jordan ML, Starzl TE, Demetris AJ. The histopathological changes associated with allograft rejection and drug toxicity in renal transplant recipients maintained on FK506. Clinical significance and comparison with cyclosporine. Am J Surg Pathol. 1993 Jan;17(1):60-8. doi: 10.1097/00000478-199301000-00007. PMID 7680544
- [Background] Birkeland SA. Steroid-free immunosuppression after kidney transplantation with antithymocyte globulin induction and cyclosporine and mycophenolate mofetil maintenance therapy. Transplantation. 1998 Nov 15;66(9):1207-10. doi: 10.1097/00007890-199811150-00016. PMID 9825819
- [Background] Calne R, Friend P, Moffatt S, Bradley A, Hale G, Firth J, Bradley J, Smith K, Waldmann H. Prope tolerance, perioperative campath 1H, and low-dose cyclosporin monotherapy in renal allograft recipients. Lancet. 1998 Jun 6;351(9117):1701-2. doi: 10.1016/S0140-6736(05)77739-4. No abstract available. PMID 9734890
- [Background] Calne RY. Initial Experience with Campath-1H in Renal Transplantation. Transplantation Reviews 2003, in press.
- [Background] Knechtle SJ, Pirsch JD, H Fechner J Jr, Becker BN, Friedl A, Colvin RB, Lebeck LK, Chin LT, Becker YT, Odorico JS, D'Alessandro AM, Kalayoglu M, Hamawy MM, Hu H, Bloom DD, Sollinger HW. Campath-1H induction plus rapamycin monotherapy for renal transplantation: results of a pilot study. Am J Transplant. 2003 Jun;3(6):722-30. doi: 10.1034/j.1600-6143.2003.00120.x. PMID 12780564
- [Background] Kirk AD, Hale DA, Mannon RB, Kleiner DE, Hoffmann SC, Kampen RL, Cendales LK, Tadaki DK, Harlan DM, Swanson SJ. Results from a human renal allograft tolerance trial evaluating the humanized CD52-specific monoclonal antibody alemtuzumab (CAMPATH-1H). Transplantation. 2003 Jul 15;76(1):120-9. doi: 10.1097/01.TP.0000071362.99021.D9. PMID 12865797
- [Background] Hricik DE, Rodriguez V, Riley J, Bryan K, Tary-Lehmann M, Greenspan N, Dejelo C, Schulak JA, Heeger PS. Enzyme linked immunosorbent spot (ELISPOT) assay for interferon-gamma independently predicts renal function in kidney transplant recipients. Am J Transplant. 2003 Jul;3(7):878-84. doi: 10.1034/j.1600-6143.2003.00132.x. PMID 12814480
- [Background] Gebauer BS, Hricik DE, Atallah A, Bryan K, Riley J, Tary-Lehmann M, Greenspan NS, Dejelo C, Boehm BO, Hering BJ, Heeger PS. Evolution of the enzyme-linked immunosorbent spot assay for post-transplant alloreactivity as a potentially useful immune monitoring tool. Am J Transplant. 2002 Oct;2(9):857-66. doi: 10.1034/j.1600-6143.2002.20908.x. PMID 12392292
- [Background] Reinsmoen NL. Cellular methods used to evaluate the immune response in transplantation. Tissue Antigens. 2002 Apr;59(4):241-50. doi: 10.1034/j.1399-0039.2002.590401.x. PMID 12135422

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were approached in the transplant clinic a Northwestern Memorial Hospital. Recruitment began April 2005 and ended April 2009.
Pre-assignment Details: Before being randomized (assigned to group) into Group 1 or Group 2, patients were screened based on inclusion/exclusion criteria (see Eligibility Criteria section). Randomization was decided before transplant surgery. Before re-randomization could begin (6 months after surgery), subjects could not be showing signs of organ rejection.
Groups:
- Group 1: Alemtuzumab + TAC (Prograf) + MMF: Receive two doses of alemtuzumab (Campath-1H, 30mg) by intravenous (IV) infusion. One dose during kidney transplant surgery and the second dose on day 2 (post-surgery) to achieve peripheral T-cell depletion. IV glucocorticoids will be given prior to Campath administration to limit cytokine release syndrome in association with this monoclonal antibody. MMF on the day of surgery and continue taking it by mouth, twice daily. TAC started on the 1st day after surgery, and then taken by mouth twice daily.
Period: Overall Study
Arm/Group | Group 1: Alemtuzumab + TAC (Prograf) + MMF | Group 2: Alemtuzumab + Sirolimus + MMF
Started | 24 (Consented:Randomized-Group 1. Given MMF prior to surgery, Alemtuzumab & TAC (Prograf) day of surgery) | 16 (Consented: Randomized-Group 2. Given Sirolimus & MMF prior to surgery, Alemtuzumab day of surgery.)
Phase 1 | 22 (Evaluated for rejection at 6months post-transplant) | 12 (Evaluated at 6 month post-transplant to potentially be weaned off Sirolimus.)
Phase 2a | 19 (Subjects who remained on Prograf at 6mo post-transplant.) | 12 (Subject who remained on Sirolimus at 6 months post-transplant.)
Phase 2b | 3 (Subjects converted to Sirolimus post-transplant.) | 0 (Subjects weaned off Sirolimus)
Phase 3 | 0 (Subjects from Phase 2b who were weaned off Sirolimus @ 12 months post-transplant.) | 0 (# weaned off Sirolimus at 12 months post-transplant.)
Completed | 22 (Completed study participation.) | 11 (Completed study participation.)
Not Completed | 2 | 5
Not completed — Death | 0 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Alemtuzumab + TAC (Prograf) + MMF: Receive two doses of alemtuzumab (Campath-1H, 30mg) by intravenous (IV) infusion. One dose during kidney transplant surgery and the second dose on day 2 (post-surgery) to achieve peripheral T-cell depletion. IV glucocorticoids will be given prior to Campath administration to limit cytokine release syndrome in association with this monoclonal antibody. MMF on the day of surgery and continue taking it by mouth, twice daily. TAC (Prograf) started on the 1st day after surgery, and then taken by mouth twice daily.
- Total: Total of all reporting groups
Arm/Group | Group 1: Alemtuzumab + TAC (Prograf) + MMF | Group 2: Alemtuzumab + Sirolimus + MMF | Total
Number analyzed (Participants) | 24 | 16 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 16 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.45833 (11.25584) | 48.125 (11.51738) | 47.125 (11.24366)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 15 | 12 | 27
Region of Enrollment [Number; unit: participants]
  United States | 24 | 16 | 40

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Biopsy-proven Acute Allograft Rejection During the First 12 Months of Transplant.
Description: The incidence of rejection is determined by the proportion of patients experiencing biopsy proven acute allograft rejection during the first 12 months post-transplant.
Time Frame: Within 12 months post kidney transplant
Population: 33 total subjects reached the 12 month participation mark.
Measure: Number; unit: Participants
Groups:
- Groups; Group 2: Evaluated for rejection of their transplanted kidney with a biopsy.
Arm/Group | Groups | Group 2
Number analyzed (Participants) | 22 | 11
Participants | 4 | 6

2. Secondary Outcome: Severity of Acute Rejection During the First 6 and 12 Months Post-transplant
Description: The diagnosis of rejection will be based on clinical symptoms and signs, laboratory tests, and confirmed by core renal allograft biopsy.
Time Frame: Months 6-12 post-transplant
Population: Study was terminated due to efficacy and there is no data was collected for this outcome measure.
Arm/Group | Group 1: Alemtuzumab + TAC (Prograf) + MMF | Group 2: Alemtuzumab + Sirolimus + MMF
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Renal Function at 12 Months Post-transplant
Description: Laboratory tests for renal function include creatinine or iothalamate glomerular filtration rate (GFR).
Time Frame: At 12 months post-transplant
Population: Study was stopped due to efficacy and no data was collected for this outcome measure.
Groups:
- Group 1; Group 2: Evaluated for rejection of their transplanted kidney with a biopsy.
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Incidence of Donor Specific Hyporesponsiveness Allowing for the Conversion to Monotherapy
Description: The proportion of subjects for both groups determine this measure: 1) Patients in tacrolimus arm who do not experience acute rejection and demonstrate evidence of donor specific hyporesonsiveness at 9 months post-transplant (those staying on TAC+MMF) or 3 months post-convertion (converted from TAC+MMF to Sirolimus+MMF) will be weaned to MMF monotherapy; 2) Those in the sirolimus+MMF arm who do not experience acute rejection and demonstrate evidence of donor specific hyporesponsiveness at 6 months post-transplant will be weaned to MMF monotherapy.
Time Frame: At 6 & 9 months post-transplant
Population: Study was stopped due to efficacy and no data was collected for this outcome measure.
Arm/Group | Group 1: Alemtuzumab + TAC (Prograf) + MMF | Group 2: Alemtuzumab + Sirolimus + MMF
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Patient and Graft Survival Rates at 6 and 12 Months Post-transplant
Time Frame: At 6 & 12 months post-transplant
Population: Study was stopped due to efficacy and no data was collected for this outcome measure.
Arm/Group | Group 1: Alemtuzumab + TAC (Prograf) + MMF | Group 2: Alemtuzumab + Sirolimus + MMF
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Group 1: Post-conversion to Sirolimus: After conversion to Sirolimus, if no rejection of transplanted kidney within 9 months post-transplant, will be weaned off Sirolimus.
Arm/Group | Group 1: Alemtuzumab + TAC + MMF | Group 2: Alemtuzumab + Sirolimus + MMF | Group 1: Post-conversion to Sirolimus
Serious Adverse Events (participants affected / at risk) | 4/24 | 4/16 | 1/3
Other Adverse Events (participants affected / at risk) | 16/24 | 14/16 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Alemtuzumab + TAC + MMF (N=24) | Group 2: Alemtuzumab + Sirolimus + MMF (N=16) | Group 1: Post-conversion to Sirolimus (N=3)
Deep vein thrombosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Pulmonary emboli (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypertension/respiratory distress post kidney biospy (Cardiac disorders) | 1 | 0 | 0
CMV (Infections and infestations) | 1 | 0 | 0
Abdominal hernia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Would dishiscence (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Community aquired pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Alemtuzumab + TAC + MMF (N=24) | Group 2: Alemtuzumab + Sirolimus + MMF (N=16) | Group 1: Post-conversion to Sirolimus (N=3)
Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Shingles (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Severe cellular rejection (Renal and urinary disorders) | 1 | 0 | 0
Antibody mediated rejection (Renal and urinary disorders) | 1 | 0 | 1
Right upper quadrant pain post conversion to rapamune (General disorders) | 1 | 0 | 0
Orthostatic hypertension (Cardiac disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 0
Pyelonephritis (Renal and urinary disorders) | 0 | 1 | 0
Hyperkalemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Bladder spasms (Renal and urinary disorders) | 1 | 0 | 0
Positive sputum culture (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Renal and urinary disorders) | 2 | 0 | 0
Nausea, vomiting, diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Cellulitis of AV fistula repair site (Infections and infestations) | 0 | 1 | 0
Fluid collection around kidney (Renal and urinary disorders) | 0 | 1 | 0
Abdominal pain (General disorders) | 0 | 2 | 0
Fever (Infections and infestations) | 4 | 3 | 0
Acute allograft rejection (Renal and urinary disorders) | 1 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No